CLINICAL TRIAL: NCT05165602
Title: Evaluation of HER2-targeted Therapy for Gastric Cancer and Establishment and Verification of Monitoring System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director, Head of gastrointestinal oncology, Principal Investigator, Clinical Professor, Peking University
Other Study IDs: 68Ga-PET
Record Dates: First submitted 2021-07-05; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: HER2 Positive Gastric Cancer
Keywords: HER2 positive gastric cancer; 68Ga-HER2-affibody PET / CT; 18F-FDG PET / CT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 8 ml of blood was collected for detection of HER2 copy number in peripheral blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The positive rate of HER2 in Chinese patients with gastric cancer is about 12-13%. HER2 positive gastric cancer has strong invasion, high metastasis rate and poor prognosis. The effective rate of chemotherapy combined with anti-HER2 targeted therapy for HER2 positive advanced gastric cancer was 47%, and the median survival time was extended to 13.8 months. However, the status of HER2 in advanced gastric cancer has obvious temporal and spatial heterogeneity, and the heterogeneity of HER2 directly affects the outcome of anti-HER2 treatment. Therefore, compared with biopsy pathology, it is urgent to explore noninvasive, systemic and repeatable methods to evaluate HER2 status of systemic lesions. 68Ga-HER2 Affibody-BCH, a HER2 imaging agent, was independently prepared by the Department of nuclear medicine of our center. According to the results of preclinical studies, in patients with HER2 positive advanced gastric cancer, the imaging effect was the best 2 hours after intravenous injection of 68Ga-HER2 Affibody and there was no adverse reaction. 68Ga-HER2 Affibody PET/CT imaging can directly reflect the HER2 heterogeneity within the same lesion and between the primary and metastatic lesions. In order to solve the clinical problems, this study intends to further explore the imaging of 68Ga-HER2 Affibody-BCH in patients with advanced gastric cancer and the amplification of HER2 in the peripheral blood of this population, so as to overcome the heterogeneity of HER2, explore the potential beneficiaries of anti HER2 treatment, and provide the basis for the evaluation of anti-HER2 treatment efficacy.

DETAILED DESCRIPTION:
1.Background China is a high incidence area of digestive tract cancer. Human epidermal growth factor receptor-2 (HER2) is a transmembrane receptor like protein that binds to cell membrane. It has tyrosine kinase activity and participates in cell growth, activation and proliferation by activating downstream signaling pathways. The positive expression of HER2 in gastric cancer was defined as pathological immunohistochemistry HER2 (3 +) or HER2 (2 +) with fish detection of gene amplification. The positive rate of HER2 in Chinese patients with gastric cancer is about 12-13% . The effective rate of chemotherapy combined with anti-HER2 targeted therapy for HER2 positive advanced gastric cancer was 47%, and the median survival time was extended to 13.8 months . However, HER2 heterogeneity directly affects the outcome of anti HER2 treatment . Therefore, compared with biopsy pathology, it is urgent to explore noninvasive, systemic and repeatable methods to evaluate HER2 status of systemic lesions. PET is the abbreviation of positron emission tomography. However, the application of 18F-FDG in tumor has some limitations, such as false positive or false negative, which can not effectively distinguish tumor and inflammation. The uptake of 18F-FDG by tumor is easily affected by pathological or physiological factors, such as local blood flow, oxygen content and necrosis . In recent years, researchers have devoted themselves to the development of new specific tumor imaging agents, among which human epidermal growth factor receptor 2 (HER2) imaging agent is a research hotspot.

Affibody, also known as "artificial antibody", is a type of engineered scaffold proteins, based on nonimmune protein affinity ligands. Compared with the antibody, the small size affibody has some unique advantages: 1) It has small molecular weight and simple structure, which could be synthesized and modified by peptide synthesizer. 2) It has high selectivity and affinity, but low nonspecific binding rate. 3) It has strong tissue permeability. Affibody quickly accumulates in the tumors and rapidly excretes from normal organs (blood, muscle etc.). And images with high contrast could be obtained only at few hours after administration. In recent years, the application of HER2 targeted affibody (ZHER2:342) and its analogues (ZHER2:2891 and ZHER2:2395) in tumor molecular imaging is beginning to attract people's attention. Gabriela Kramer-Marek compared the imaging performance of 18F-FBEM-cys-ZHER2:342 and 18F-FDG in nude mice with MDA-MB-231 tumor and lung metastasis. 18F-FBEM-cys-ZHER2:342 successfully targeted HER2 positive lung metastases, while 18F-FDG not detected metastasis for the interfered by peripheral inflammation and normal tissues.

68Ga is a new type of positron nuclide, which is produced by 68Ge-68Ga generator. The mother nuclide 68Ge is a long-lived radioisotope with a half-life of 271 days, which can be stored in the generator for about one year.

68Ga is easy to obtain, and the high purity 68Ga can be refresh after 4 hours, which is conducive to multi imaging on the same day. The physical half-life of 68Ga is 68 min, and 89% of the decay process is positron decay, Emax is 1.92 MeV, and the remaining 11% is electron capture. Compared with cyclotron, 68Ge-68Ga generator is in small size, does not need special site with radiation shielding structure, and has lower requirements for equipment operation and maintenance personnel. Compared with 18F, 68Ga has the advantages of low cost, simple preparation and fast labeling. Therefore, 68Ga labeled HER2 affinity probe is of great significance for in vivo monitoring of HER2 status. The 68Ga labeled affinity probe 68Ga-ABY-002 (68Ga-DOTA-ZHER2:342-pep) was prepared by Uppsala University in Sweden. The result showed that 68Ga-ABY-002 successfully detected lung metastases from breast cancer. However, there was no good detection effect of liver metastases for high uptake of the normal abdominal tissue, especially the liver background.

2 .The Work and Conditions of Our Center 68Ga-HER2-affibody-BCH was prepared by the department of nuclear medicine of Peking University Cancer Hospital. The time is only 30 minutes and the yield is 80% ± 5%. The radiochemical purity was more than 95%. Micro-PET imaging showed high uptake in tumors with ovarian cancer and breast cancer. In view of the convenient synthesis and good imaging performance, 68Ga-HER2-affibody-BCH is expected to be widely used in clinical diagnosis, differentiation and efficacy detection of HER2 positive tumors.

3.Bio-distribution and Imaging of 68Ga-HER2-affibody-BCH in Models

1. Bio-distribution of 68Ga-HER2-affibody-BCH in normal mice Normal ICR mice (20-25 g) were randomly divided into 7 groups with 6 mice in each group, half male and half female. The mice were anesthetized with isoflurane (2-3%). Injected with 1.66 MBq 68Ga-HER2-affibody-BCH (0.2 ml) via tail vein. Then the mice were killed at different time points (5, 10, 30, 60, 90, 120, 240 min) after injection. The organs of interest were dissected and taken out. The radioactivity and weight of each organ were measured with gamma counter, and the radioactivity percentage per unit mass of organ was calculated.

   The bio-distribution study of 68Ga-HER2-affibody-BCH in normal mice showed: 68Ga-HER2-affibody-BCH was rapidly cleared, and the radioactivity in blood was only 0.27 %ID/g after 120 min injection. The uptake of 68Ga-HER2-affibody-BCH in kidney was high, suggesting that the probe was excreted mainly through urinary system; The probe had low uptake in the liver, and the metabolic rate was fast; The initial brain uptake was only 0.87 %ID/g. The initial uptake of radioactivity in bone was low and decreased with the injection time, which indicated that 68Ga-HER2-affibody-BCH was stable in vivo. In the course of animal bio-distribution study, the vital signs and behaviors of all mice did not change significantly.
2. Micro-PET Imaging of 68Ga-HER2-affibody-BCH in PDX Models of Gastric Cancer PDX model is known as "the living specimen bank of patients' specimen renewable". Prof. Shen and her team established the best large-scale advanced gastric cancer PDX model library for preclinical research for the first time. Preliminary results show that PDX model has unique advantages in micro-PET imaging with 68Ga-HER2-affibody-BCH.

4.Preliminary exploration of 68Ga-HER2-affibody-BCH in patients with gastric cancer According to the results of preclinical research, 68Ga-HER2-affibody has been approved by the Ethics Committee (approval No. 2018kt61) and has been initially applied in HER2 imaging of patients with advanced gastric cancer. Previous results showed that in HER2 positive patients with advanced gastric cancer, 68Ga-HER2-affibody was effective 2 hours after intravenous injection,The result was the best, and there was no adverse reaction. 68Ga-HER2-affibody PET / CT imaging can directly reflect the HER2 heterogeneity within the same lesion and between the primary and metastatic lesions. In 13 HER2 negative patients, 2 patients showed positive 68Ga-HER2-affibody PET / CT imaging, and 2 patients had certain benefits after anti-HER2 treatment. Among them, 68Ga-HER2-affibody is more sensitive than 18F-FDG, which is not sensitive to signet ring cell carcinoma / Lauren type diffuse gastric cancer imaging. In addition, four HER2 positive patients underwent dynamic monitoring during treatment. The results showed that 68Ga-HER2-affibody PET / CT could clearly show peritoneal nodules in patients with peritoneal metastasis without RECIST standard target lesions. At the same time, it was observed that the dynamic changes of 68Ga-HER2-affibody SUVmax before and after treatment were related to the response to anti-HER2 treatment.

5.

1. Objective: To compare the diagnostic efficacy of 68Ga-HER2-affibody and 18F-FDG in the malignant differentiation and staging of HER2 positive tumor patients, and to further explore the imaging of 68Ga-HER2-affibody PET/ CT in patients with advanced gastric cancer and the amplification of HER2 in peripheral blood of this population, so as to overcome the heterogeneity of HER2 and explore the potential beneficiaries of anti HER2 therapy, At the same time, it provides the basis for the evaluation of anti HER2 treatment.
2. Significance: The most commonly used tumor imaging agent of pet is 18F-deoxyglucose (18F-FDG), which reflects the glucose metabolism of tumor cells. However, its application in tumor has some defects. The uptake of 18F-FDG by tumor is easily affected by pathological or physiological factors such as local blood flow, oxygen content and necrosis. In recent years, researchers are committed to the development of new specific tumor imaging agents, in order to improve the diagnostic rate of tumor. Human epidermal growth factor receptor 2 (HER2) imaging agent is a research hotspot. Human epidermal growth factor receptor-2 (HER2) is a transmembrane receptor like protein that binds to cell membrane. It has tyrosine kinase activity and participates in cell growth, activation and proliferation by activating downstream signaling pathways. Studies have shown that HER2 is not expressed in normal tissues, but it is highly expressed in breast cancer, gastric cancer, cervical cancer and other malignant tumors. It is one of the specific targets of tumor diagnosis and treatment. This project provides a clinically available PET molecular probe 68Ga-HER2-affibody BCH targeting HER2 to improve the accuracy of tumor diagnosis and individualized treatment。 6.Implementation plan 6.1 Trial design: single center, randomized, open, self-control study. 6.2 Case selection criteria: 1) unresectable or metastatic adenocarcinoma of the gastroesophageal junction confirmed by pathology and imaging; 2) Subjects had measurable lesions according to recist1.1, or unmeasurable but evaluable lesions; 3) HER2 (1 +) or HER2 (2 +) or HER2 (3 +) was found in primary or metastatic lesions; 4) Age: over 18 years old; 5) ECOG was 0-2; 6) Voluntary participation and written informed consent; exclusion criteria: 1) The inclusion criteria were not met; 2) The function of liver and kidney was abnormal; 3) Cardiac insufficiency; 4) Preparation of pregnant, pregnant and lactating women; 5) Unable to lie on your back for 30 minutes; 6) Those who refused to join the clinical study; 7) Those who have no legal capacity or whose medical or ethical reasons affect the continuation of the research; 8) Refuse to provide tissue or hematological samples.

6.3 Sample size and dosage: from March 2021 to March 2023, 30 subjects will be included. All subjects were required to receive 18F-FDG and 68ga-her2affibody BCH intravenous injection, and PET / CT imaging within the specified time.

6.4 Test process:

1. The patients were screened, 68Ga-HER2-affibody PET/ CT was completed, 18F-FDG PET / CT imaging was performed on different days within one week, and 8 ml blood was taken to detect the copy number of HER2 in peripheral blood;
2. Patients with 68Ga-HER2-affibody PET / CT positive lesions or peripheral blood HER2 copy number positive lesions were included;
3. After treatment, the efficacy was evaluated every 6 cycles;
4. 68Ga-HER2-affibody PET / CT and the copy number of HER2 in peripheral blood were reexamined 6 weeks after treatment;
5. After confirming the progress of treatment, 68Ga-HER2-affibody PET/ CT and the copy number of HER2 in peripheral blood were checked again;
6. Radionuclide images of patients were collected to establish a prediction model. The consistency and difference of HER2 expression with 68Ga-HER2-affibody PET / CT and HER2 copy number expression in peripheral blood were evaluated. The correlation between the efficacy of anti-HER2 treatment and the dynamic changes of 68Ga-HER2-affibody PET / CT expression was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. unresectable or metastatic adenocarcinoma of the gastroesophageal junction confirmed by pathology and imaging;
2. Subjects had measurable lesions according to recist1.1, or unmeasurable but evaluable lesions;
3. HER2 (1 +) or HER2 (2 +) or HER2 (3 +) was found in primary or metastatic lesions;
4. Age: over 18 years old;
5. ECOG was 0-2;
6. Voluntary participation and written informed consent;

Exclusion Criteria:

1. The inclusion criteria were not met;
2. The function of liver and kidney was abnormal;
3. Cardiac insufficiency;
4. Preparation of pregnant, pregnant and lactating women;
5. Unable to lie on your back for 30 minutes;
6. Those who refused to join the clinical study;
7. Those who have no legal capacity or whose medical or ethical reasons affect the continuation of the research;
8. Refuse to provide tissue or hematological samples. 9）Allergic to both of the contrast agents used in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with high HER2 expression in gastric / gastroesophageal junction adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
the relationship between 68Ga SUVmax before treatment and the therapeutic effect will be assessed by SPSS26.0 | 3 years
  The 68Ga SUVmax lesion will be determined by nuclear medicine doctors, and the efficacy will be determined according to Resist1.1 by physicians.Then SPSS 26.0 will be used to analyze the relationship between the two.

SECONDARY OUTCOMES:
the relationship between the dynamic change of 68Ga SUVmax and the therapeutic effect will be assessed by SPSS26.0 | 3 years
  The dynamic change of 68Ga SUVmax will be determined by nuclear medicine doctors, and the efficacy will be determined according to Resist1.1 by physicians.Then SPSS 26.0 will be used to analyze the relationship between the two.

CONTACTS AND LOCATIONS:
Overall Officials: lin shen, Professor, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Wang J, Xu R, Li J, Bai Y, Liu T, Jiao S, Dai G, Xu J, Liu Y, Fan N, Shu Y, Ba Y, Ma D, Qin S, Zheng L, Chen W, Shen L. Randomized multicenter phase III study of a modified docetaxel and cisplatin plus fluorouracil regimen compared with cisplatin and fluorouracil as first-line therapy for advanced or locally recurrent gastric cancer. Gastric Cancer. 2016 Jan;19(1):234-44. doi: 10.1007/s10120-015-0457-4. Epub 2015 Jan 21. PMID 25604851
- [Background] Lu Z, Zhang X, Liu W, Liu T, Hu B, Li W, Fan Q, Xu J, Xu N, Bai Y, Pan Y, Xu Q, Bai W, Xia L, Gao Y, Wang W, Shu Y, Shen L. A multicenter, randomized trial comparing efficacy and safety of paclitaxel/capecitabine and cisplatin/capecitabine in advanced gastric cancer. Gastric Cancer. 2018 Sep;21(5):782-791. doi: 10.1007/s10120-018-0809-y. Epub 2018 Feb 27. PMID 29488121
- [Background] Van Cutsem E, Bang YJ, Feng-Yi F, Xu JM, Lee KW, Jiao SC, Chong JL, Lopez-Sanchez RI, Price T, Gladkov O, Stoss O, Hill J, Ng V, Lehle M, Thomas M, Kiermaier A, Ruschoff J. HER2 screening data from ToGA: targeting HER2 in gastric and gastroesophageal junction cancer. Gastric Cancer. 2015 Jul;18(3):476-84. doi: 10.1007/s10120-014-0402-y. Epub 2014 Jul 20. PMID 25038874
- [Background] Sheng WQ, Huang D, Ying JM, Lu N, Wu HM, Liu YH, Liu JP, Bu H, Zhou XY, Du X. HER2 status in gastric cancers: a retrospective analysis from four Chinese representative clinical centers and assessment of its prognostic significance. Ann Oncol. 2013 Sep;24(9):2360-4. doi: 10.1093/annonc/mdt232. Epub 2013 Jun 19. PMID 23788757
- [Background] Huang D, Lu N, Fan Q, Sheng W, Bu H, Jin X, Li G, Liu Y, Li X, Sun W, Zhang H, Li X, Zhou Z, Yan M, Wang X, Sha W, Ji J, Cheng X, Zhou Z, Xu J, Du X. HER2 status in gastric and gastroesophageal junction cancer assessed by local and central laboratories: Chinese results of the HER-EAGLE study. PLoS One. 2013 Nov 14;8(11):e80290. doi: 10.1371/journal.pone.0080290. eCollection 2013. PMID 24244671
- [Background] Qiu M, Zhou Y, Zhang X, Wang Z, Wang F, Shao J, Lu J, Jin Y, Wei X, Zhang D, Wang F, Li Y, Yang D, Xu R. Lauren classification combined with HER2 status is a better prognostic factor in Chinese gastric cancer patients. BMC Cancer. 2014 Nov 7;14:823. doi: 10.1186/1471-2407-14-823. PMID 25380654
- [Background] Bao W, Fu HJ, Xie QS, Wang L, Zhang R, Guo ZY, Zhao J, Meng YL, Ren XL, Wang T, Li Q, Jin BQ, Yao LB, Wang RA, Fan DM, Chen SY, Jia LT, Yang AG. HER2 interacts with CD44 to up-regulate CXCR4 via epigenetic silencing of microRNA-139 in gastric cancer cells. Gastroenterology. 2011 Dec;141(6):2076-2087.e6. doi: 10.1053/j.gastro.2011.08.050. Epub 2011 Sep 16. PMID 21925125
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Park SR, Park YS, Ryu MH, Ryoo BY, Woo CG, Jung HY, Lee JH, Lee GH, Kang YK. Extra-gain of HER2-positive cases through HER2 reassessment in primary and metastatic sites in advanced gastric cancer with initially HER2-negative primary tumours: Results of GASTric cancer HER2 reassessment study 1 (GASTHER1). Eur J Cancer. 2016 Jan;53:42-50. doi: 10.1016/j.ejca.2015.09.018. Epub 2015 Dec 13. PMID 26693898
- [Background] Ahn S, Ahn S, Van Vrancken M, Lee M, Ha SY, Lee H, Min BH, Lee JH, Kim JJ, Choi S, Jung SH, Choi MG, Lee JH, Sohn TS, Bae JM, Kim S, Kim KM. Ideal number of biopsy tumor fragments for predicting HER2 status in gastric carcinoma resection specimens. Oncotarget. 2015 Nov 10;6(35):38372-80. doi: 10.18632/oncotarget.5368. PMID 26460823
- [Background] Yagi S, Wakatsuki T, Yamamoto N, Chin K, Takahari D, Ogura M, Ichimura T, Nakayama I, Osumi H, Shinozaki E, Suenaga M, Fujisaki J, Ishikawa Y, Yamaguchi K, Namikawa K, Horiuchi Y. Clinical significance of intratumoral HER2 heterogeneity on trastuzumab efficacy using endoscopic biopsy specimens in patients with advanced HER2 positive gastric cancer. Gastric Cancer. 2019 May;22(3):518-525. doi: 10.1007/s10120-018-0887-x. Epub 2018 Oct 17. PMID 30328533
- [Background] Kramer-Marek G, Bernardo M, Kiesewetter DO, Bagci U, Kuban M, Aras O, Zielinski R, Seidel J, Choyke P, Capala J. PET of HER2-positive pulmonary metastases with 18F-ZHER2:342 affibody in a murine model of breast cancer: comparison with 18F-FDG. J Nucl Med. 2012 Jun;53(6):939-46. doi: 10.2967/jnumed.111.100354. Epub 2012 May 11. PMID 22582046
- [Background] Velikyan I. 68Ga-Based radiopharmaceuticals: production and application relationship. Molecules. 2015 Jul 16;20(7):12913-43. doi: 10.3390/molecules200712913. PMID 26193247